CLINICAL TRIAL: NCT05080101
Title: Effect Sof Basic Body Awareness Therapy on Posture, Pain, Disability, Quality of Life, Sleep Quality and Body Awareness in Individual With Chronic Low Back Pain
Brief Title: Effects of Basic Body Awareness Therapy on Pain, Sleep, Disability and Quality of Life in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kaniye Üneş, PT, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020/14-11 (KA-20021)
Record Dates: First submitted 2021-10-02; First posted 2021-10-15 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Chronic Low-back Pain
Keywords: Pain; Quality of Life; Disability; Sleep; Body Awareness
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: A total of 28 individual diagnosed with chronic low back pain will be included in this study. The patients who meet the inclusion criteria will be divided into 2 groups randomly as study (n=14) and control (n=14). Patients in control group will receive 40-mins conventional physiotherapy session for 3-days per week, over 6 weeks. Conventional physiotherapy will consist of stretching and strengthening exercises, postural alignment exercises, as well as electrotherapy such as transcutaneous electric magnetic stimulation. Patients in study group will receive Basic Body Awareness Therapy (BBAT) 3 days in a week, over 6 weeks in addition to conventional physiotherapy. BBAT will consist of flexibility exercises and cognitive exercises
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physiotherapy Group (Active Comparator): Patients in control group (n=14) will receive 40-mins conventional physiotherapy session for 3-days per week, over 6 weeks. Conventional physiotherapy will consist of stretching and strengthening exercises, postural alignment exercises, as well as electrotherapy such as transcutaneous electric magnetic stimulation (TENS) which will be applied to lumbar region with a frequency of 100 Hz, 50-100 μsec current duration for 20 minutes, hotpack which will be applied to lumbar region for 20 mins, and ultrasound application which will be applied to the lumbar region with a Chattanooga Intelect Mobile device at a frequency of 1 MHz, at a dose of 1.5 W/cm2, for 6 minutes using a 10 cm2 head.
  Interventions: Other: Conventional Therapy Program
- Basic Body Awareness Therapy Group (Experimental): Patients in study group (n=14) will receive Basic Body Awareness Therapy (BBAT) 3 days in a week, over 6 weeks in addition to conventional physiotherapy. BBAT will consist of flexibility exercises and various cognitive exercises in supine, position, sitting position and standing position. These exercises will be consist of exercises such as body scanning, breathing, sound resonance.
  Interventions: Other: Basic Body Awareness Therapy Group Program

INTERVENTIONS:
Other: Conventional Therapy Program — Patients in control group (n=14) will receive 40-mins conventional physiotherapy session for 3-days per week, over 6 weeks. Conventional physiotherapy will consist of stretching and strengthening exercises, postural alignment exercises, as well as electrotherapy such as transcutaneous electric magnetic stimulation (TENS) which will be applied to lumbar region with a frequency of 100 Hz, 50-100 μsec current duration for 20 minutes, hotpack which will be applied to lumbar region for 20 mins, and ultrasound application which will be applied to the lumbar region with a Chattanooga Intelect Mobile device at a frequency of 1 MHz, at a dose of 1.5 W/cm2, for 6 minutes using a 10 cm2 head.
  Arms: Conventional Physiotherapy Group
Other: Basic Body Awareness Therapy Group Program — Patients in study group (n=14) will receive Basic Body Awareness Therapy (BBAT) 3 days in a week, over 6 weeks in addition to conventional physiotherapy. BBAT will consist of flexibility exercises and various cognitive exercises in supine, position, sitting position and standing position. These exercises will be consist of exercises such as body scanning, breathing, sound resonance.
  Arms: Basic Body Awareness Therapy Group

SUMMARY:
Chronic low back pain is a common problem worldwide. In treatment, conservative methods usually are used. Basic Body Awareness Therapy is related to mindfulness-based therapies and meditation techniques. It is a method that has been used and found effective in some diseases affecting the musculoskeletal system. Therefore, in this study, body awareness was applied in addition to conventional treatment in patients with chronic low back pain.

DETAILED DESCRIPTION:
Throughout a lifetime, chronic low back pain is a common problem that affects approximately 80% of people. Among musculoskeletal system problems, it is one of the most commonly observed issues. There are various treatment methods available. The absence of evidence-based treatment guidelines negatively affects the choice of treatment to be applied. There are medical and conservative treatment options. These methods include acupuncture, transcutaneous electrical nerve stimulation, injection therapy, non-steroidal anti-inflammatory drugs, and lumbar supports. Basic Body Awareness Therapy is a physiotherapy treatment method that has been developed in the Scandinavian countries over the course of the last two decades. This innovative approach focuses on enhancing body awareness and has gained recognition as an effective therapeutic technique in the field of physiotherapy. Basic Body Awareness Therapy has been applied as a secondary treatment method in various conditions such as fibromyalgia, neck pain, and ankylosing spondylitis, and has been found to be effective. It has yielded positive results when used in addition to conventional treatments for musculoskeletal problems, as demonstrated in the literature. This study aims to apply Basic Body Awareness Therapy to individuals with chronic low back pain, based on its effectiveness in musculoskeletal issues, and create a new treatment combination. Twenty-eight patients were included in the study, and in addition to the standard treatment protocol, Basic Body Awareness Therapy exercises were administered.

ELIGIBILITY:
Inclusion Criteria:

* Having low back pain for 3 months or more
* Being between the ages of 18-65
* Not having received any back-related treatment before
* Volunteer to participate in the study

Exclusion Criteria:

* Pregnancy
* History of tumor / metastatic disease
* History of spinal trauma, spinal cord injury
* History of infection
* Presence of congenital deformity in the spine
* History of previous spinal surgery
* Having a neurological disease (Alzheimer's, Amyotrophic Lateral Sclerosis, Multiple Sclerosis, Parkinson's, Stroke)
* Having musculoskeletal problems other than low back pain (rheumatoid arthritis, pathological fractures, avascular necrosis or osteonecrosis, severe osteoarthritis, spondylo-arthropathy)
* Patients who received a physiotherapy rehabilitation program in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index Score | 5 mins
  The Oswestry Disability Index (ODI) is the gold standard, valid and reliable outcome measurement tool for assessing functionality in patients with low back pain. For 10 different functional activities, there are 6 different answers for which the patient does not know the score equivalent. Each activity is scored between 0 (functional level adequate) and 5 (severe limitation). The measurement result is expressed over the total score and the ratio of the score to the total maximum score is determined as a percentage. 0-20% minimal disability, 21-40% moderate disability, 41-60% severe disability, 61-80% bedridden, 81-100% completely bedridden or interpreted as exaggerating their situation. The minimal clinical significance level is accepted as 10%, changes occurring less than this rate are considered as measurement error.
Functional Rating Index Score | 5 mins
  The Functional Rating Index (FRI) is a valid and reliable method that evaluates the functionality and the decrease in functions caused by low back pain. FRI evaluates the functional level in 10 different domain (sleep, personal care, travel, work, etc.) that may be affected due to low back pain. FRI is a scale in which each item is scored between 0 (no pain, no restriction while doing the activity) and 4 (totally dependent, need someone else's help). Maximum score of FRI is 40 which indicates that the patient can easily perform functional activities.
New York Posture Analysis Score | 5 mins
  The New York Posture Analysis (NYPA) will be used to assess patients' posture. NYPA consists of 13 items that evaluate the static posture of the body from the lateral and posterior aspects, and each item is given a score of five (5) if the person has a correct posture, three (3) if the posture is moderately impaired, and one (1) point if there is a severe deterioration. . The posture score that the patient will receive is one of 25 different scores ranging from 13 to 65, and a higher score indicates better posture. Standard evaluation criteria developed for this test were determined as "very good" if the total score is ≥45, "good" if 40-44, "moderate" if 30-39, "poor" if 20-29, and "poor" if ≤19.
Pain Level assessed by McGill Pain Scale | 5 mins
  The McGill Pain Scale Short Form, which is a valid and reliable method used to evaluate pain, consists of three parts. In the first part, there are 15 descriptive word groups. Of these, 11 evaluate the sensory dimension of the pain, and 4 evaluate the perceptual dimension. These descriptors are rated on an intensity scale from 0 to 3 (0= none, 1= Mild, 2=Moderate, 3= Excess). In the first part of the scale, a total of 3 pain scores are obtained: sensory pain score, perceptual pain score and total pain score. In the second part of the form, there were five word groups ranging from "mild pain" to "unbearable pain" to determine the severity of the patient's pain. In the third part, the current pain intensity of the patient was evaluated using a visual comparison scale.
Sleep Quality assessed by Pittsburgh Sleep Quality Index | 5 mins
  Sleep quality of patients will be evaluated using the Pittsburgh Sleep Quality Index (PSQI), a valid and reliable assessment tool. The PSQI consists of 7 components that assess subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and loss of daytime functionality. Some of the components consist of a single item, while others consist of groupings of several items. Each item is evaluated between 0 and 3 points. It is accepted that a total scale score of 5 and above indicates poor sleep quality. The sum of these 7 component scores gives the overall index score. The total score is between 0-21. A high total score indicates poor sleep quality.
Quality of Life assessed by Short Form-12 | 5 mins
  The Health Scale Short Form-12 (SF-12), which is a valid and reliable tool, will be used to assess patients' quality of life. The SF-12 scale evaluates 8 sub-dimensions as physical function, physical role difficulty, social function, pain, mental health, emotional role difficulty, vitality, general perception of health, and 2 areas, mental health and physical health, which is a combination of these dimensions. Considering the last month, the patient scores some of the items between 1 and 3, some of them between 1 and 5, and the sum of the scores for 8 sub-dimensions and 2 domains separately is expressed as %. A higher percentage indicates a better quality of life.
Beck Depression Inventory Score | 5 mins
  Beck Depression Inventory (BDI) will be used to evaluate the depression status of the patients. BDI is a valid and reliable scale with 21 items, each of which can be scored between 0 (minimal) and 3 (severe hopelessness). The patient answers this scale himself, thinking about the last week. The sum of the scores of the items represents the scale score, and this score ranges from 0 to 63. 0-9 points are interpreted as minimal depression, 10-16 points as mild depression, 17-29 points as moderate depression and 30-63 points as severe depression.
The Body Awareness Scale Score | 5 mins
  Body Awareness Questionnaire is a valid and reliable scale that measures body awareness of individuals for different situations (illness, cold, change in energy level, etc.). It consists of a total of 18 items, each of which can be scored between 1 (completely true for me) and 7 (not true for me at all).
The Awareness: Body Chart Score | 5 mins
  The Awareness: Body Chart (ABC) is a newly developed, valid and reliable scale used to evaluate individuals' body awareness. ABC divides the human body into 51 separate regions and grades each of them separately. It does this by painting with colors, not by grading with numbers. In this coloring, orange is interpreted as "I can perceive in great detail", yellow as "I can perceive clearly", green as "I can perceive", blue as "I can perceive vaguely" and black as "I cannot perceive". The evaluator then converts these colors to numerical values from 5 to 1, respectively (for example, orange = 5). If the patient feels pain using a red felt-tip pen, he marks the area and rates the pain intensity between 0 and 100. A high ABC score of the patient means good awareness, while a high pain score means severe pain.
Body Image Questionnaire Score | 5 mins
  Body Image Questionnaire (BIQ) is a scale that determines satisfaction with one's body parts or functions. Hovardaoğlu et al. found that the scale was valid and reliable. demonstrated in the study by The scale consists of a total of 40 different items, and each item is scored between 1 (I quite like it) and 5 (I don't like it at all). A low score means that the person is satisfied with their body and functions.
Fremantle Back Awareness Questionnaire Score | 5 mins
  The Fremantle Back Awareness Questionnaire (FBAQ) is the only known valid and reliable awareness scale specific to the waist area. This scale consists of 9 items assessing denial-like symptoms, decreased proprioception, perceived body shape and size, and each item is scored between 0 (never) and 4 (always). High scores indicate decreased awareness.

CONTACTS AND LOCATIONS:
Overall Officials: Kaniye Unes, PT, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No